CLINICAL TRIAL: NCT05419440
Title: Laparoscopic Drainage Versus Interventional Radiology In Management Of Appendicular Abscess : A Randomized Controlled Trial.
Brief Title: Laparoscopic Drainage Versus Interventional Radiology In Management Of Appendicular Abscess :
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: General Surgery Departement
Record Dates: First submitted 2022-06-09; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Acute Abdomen
Keywords: appendicular abscess , laparoscopy
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled clinical trial included all patients who developed the manifestations of appendicular abscess and referred to the Zagazig University Hospital Emergency Department between January 2020 and February 2022. The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 55342/24.1.2020), The sample size was 172 patients divided into two equal group group (1) laparoscopic group involved 86 patients & group (2) interventional radiology group involved 86 patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic drainage of appendicular abscess (Active Comparator): laparoscopic drainage of appendicular abscess laparoscopy drainage of pus ,excision of appendix and putting a drain
  Interventions: Procedure: laparoscopic drainage of appendicular abscess
- interventional radiology for management of appendicular abscess (No Intervention): insertion of a drain or pig tail under sonar or ct guided

INTERVENTIONS:
Procedure: laparoscopic drainage of appendicular abscess — access to caecum and remove any adhesions with surrounding by sharp & blunt dissection , then access to appendicular abscess by sharp and blunt dissection after complete separation of the appendix from surrounding & complete drainage of pus & removal of all necrotic tissue , removal of the remnant appendix , in cases with healthy base of appendix ,we closed the stump with endo-loop , in case with unhealthy base , we closed the stump by suturing by ethibond 2/0 in two layers in case with little edema & inflammation of caecum ( sutures not cut through ) , in cases with marked edema and inflammation of caecum , we close the site of base by omental patch fixed by taking full thickness sutures in wall of caecum and pass through omental patch , we examine any leak by pressing on caecum and observe any fecal matter comes & air leak test , in all cases we put large drain at pelvis
  Arms: laparoscopic drainage of appendicular abscess

SUMMARY:
This prospective randomized controlled clinical trial included all patients who developed the manifestations of appendicular abscess and referred to the Zagazig University Hospital Emergency Department between January 2020 and February 2022. The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 55342/24.1.2020). The sample size was 172 patients divided into two equal group group (1) laparoscopic group involved 86 patients & group (2) interventional radiology group involved 86 patients.

DETAILED DESCRIPTION:
This prospective randomized controlled clinical trial included all patients who developed the manifestations of appendicular abscess and referred to the Zagazig University Hospital Emergency Department between January 2020 and February 2022. The study was prospectively approved by Zagazig University Faculty of Medicine Institutional Review Board (Approval Number: 55342/24.1.2020), and was retrospectively submitted in clinicaltrials.gov in September 2021 (NCT05051683). The study was performed in accordance with the code of ethics of the World Medical Association (Declaration of Helsinki) for studies involving human subjects. Written informed consent was obtained from all participants after explaining to them all the study procedures with its benefits and hazards. Patients ≥16- ≤60 years-old, with appendicular abscess , with early sepsis , no septic shock , ASA I & II , no other pathology and candidate for laparoscopy were deemed eligible for randomization. We excluded patients who were <16- >60 years-old, septic shock, appendicular mass, ASA III , previous abdominal operations, immune compromised patients , patients with immune suppressive therapy, pregnant patients and not candidate for laparoscopy.

Involved patients were simply randomized at a 1:1 ratio to "laparoscopic Group (LG)" or "Interventional Radiology Group (IG)" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the procedure.

The sample size was calculated by using open Epi program depending on the following data ; confidence interval 95%, power of the test 80%, ratio of unexposed/exposed 1, percent of patients with complications after management of appendicular abscess by interventional radiology 15 %, and those managed by laparoscopy 2 % , odds ratio 8.7 , and risk ratio 7.5, So the calculated sample size equal 172 patients divided into two equal group.

Primary and secondary outcomes were fecal fistula , recurrent collection and quality of life in each group after the procedures during the 3-months follow-up period, respectively.

Diagnosis After full history taking ( throbbing pain at right iliac fossa several days ago ) and complete physical examination ( fluctuant high grade fever especially at evening , severe pain & tenderness at right iliac fossa , toxic manifestations), appendicular abscess was clinically suspected and then confirmed by laboratory investigations (complete blood picture (WBC count more than 16000), liver and kidney functions, coagulation profile), radiological imaging (abdominal US or CT abdomen with oral and I.V contrast confirms appendicular abscess) , in laparoscopic group we exclude patients with other pathology after laparoscopic exploration However, the radiology finding was consistent with appendicular abscess.

Intervention For laparoscopic group ( included 86 patients ) , the patients were subjected to the following steps after the diagnosis has been confirmed as appendicular abscess. The patients were taken rapidly to operative theater , general anesthesia was given , patients were put in supine position , sterilization of the abdomen from subcostal margin to pubic bone was done , ports insertion was done , one 10 mm port supra-umbilical , one 5mm port at left iliac fossa , one 5mm port at right iliac fossa , insertion of the 10 mm port was done first by open method or versus needle , insufflation of co2 up to 14 mm.hg was done after 10 mm port insertion , exploration of the abdomen first by 10 mm telescope , to exclude other pathology and confirm the diagnosis ( we exclude patients with other pathology after laparoscopic exploration ) , then insertion of other two ports under vision , removal of any adhesions first , irrigation & suction whole the abdomen first with warm saline 0.9% , access to caecum by tilting the table head down and to left to pull all intestine away from caecum , access to caecum and remove any adhesions with surrounding by sharp & blunt dissection , then access to appendicular abscess by sharp and blunt dissection , drain all the pus by suction , irrigation with warm saline , after complete separation of the appendix from surrounding & complete drainage of pus & removal of all necrotic tissue , removal of the remnant appendix , in cases with healthy base of appendix ,we closed the stump with endo-loop , in case with unhealthy base , we closed the stump by suturing by ethibond 2/0 in two layers in case with little edema & inflammation of caecum ( sutures not cut through ) , in cases with marked edema and inflammation of caecum , we close the site of base by omental patch fixed by taking full thickness sutures in wall of caecum and pass through omental patch , we examine any leak by pressing on caecum and observe any fecal matter comes & air leak test , in all cases we made irrigation & suction with 2000cc warm saline and put large drain at pelvis to be removed later according to its discharge , deflation of the abdomen and close the port sites. Then patients were kept in hospital under observation till drain removal.

For interventional radiology group ( included 86 patients ) , patients were subjected for drain insertion or pig catheter insertion at right iliac fossa under a complete sterilized filed by radiologist , then daily wash from drain or pig catheter by gentamycin & metronidazole till drain discharge comes clear fluid , then drain removed according the amount of discharge and doing us confirm there is no residual.

Statistical analysis Analysis of data was performed using SPSS (Statistical Package of Social Services) version 22. Quantitative variables were described as mean (±SD, standard deviation) and median (range) according to Shapiro test of normality. Qualitative variables were described as a number and a percent. Chi-square test was used to compare qualitative variables between the 2 groups. Fisher exact test was used when one expected cell or more are less than 5. Unpaired t-test was used to compare quantitative variables, in parametric data (SD < 30% of the mean). Mann Whitney test was used instead of unpaired t-test in non-parametric data (SD > 30% of the mean). The results were considered statistically significant when the significant probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically significant (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥16- ≤60 years-old with appendicular abscess
* with early sepsis.
* no septic shock.
* ASA I & II.
* no other pathology .
* candidate for laparoscopy .

Exclusion Criteria:

* <16- >60 years-old .
* septic shock.
* appendicular mass.

  *, ASA III .
* previous abdominal operations.
* immune compromised patients .
* patients with immune suppressive therapy.
* pregnant patients not
* candidate for laparoscopy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
incidence of complications after laparoscopic drainage of appendicular abscess | within one week after laparoscopic drainage of the appendicular abscess
  incidence of complications after laparoscopic drainage of appendicular abscess

SECONDARY OUTCOMES:
incidence of mortality after laparoscopic drainage of appendicular abscess | within one month after laparoscopic drainage of appendicular abscess
  incidence of mortality after laparoscopic drainage of appendicular abscess

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — Zagazig University Hospitals
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharquia, Egypt

IPD SHARING:
Plan to Share IPD: No